CLINICAL TRIAL: NCT05013983
Title: Single-center, Randomized, Double-blind, Placebo-controlled Phase I/II Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of Recombinant COVID-19 Vaccine (Sf9 Cells) in Healthy People Aged 6-17 Years
Brief Title: Clinical Trial of Recombinant COVID-19 Vaccine (Sf9 Cells) in Children and Adolescents
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Clinical trials not conducted
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT125
Record Dates: First submitted 2021-08-17; First posted 2021-08-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
Keywords: Safety; Immunogenicity; COVID-19 Vaccine; Recombinant vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Low-dose vaccine (6-11 years) (Experimental): three doses of low-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21，42.
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cells)
- Medium-dose vaccine (6-11 years) (Experimental): three doses of medium-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21，42.
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cells)
- Medium-dose vaccine (12-17 years) (Experimental): three doses of medium-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21，42.
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cells)
- High-dose vaccine (12-17 years) (Experimental): three doses of high-dose Recombinant COVID-19 vaccine (Sf9 cells) at the schedule of day 0, 21，42.
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cells)
- Low-dose placebo (6-11 years) (Placebo Comparator): three doses of low-dose placebo at the schedule of day 0, 21，42.
  Interventions: Other: Placebo control
- Medium-dose placebo (6-11 years) (Placebo Comparator): three doses of medium-dose placebo at the schedule of day 0, 21，42.
  Interventions: Other: Placebo control
- Medium-dose placebo (12-17 years) (Placebo Comparator): three doses of medium-dose placebo at the schedule of day 0, 21，42.
  Interventions: Other: Placebo control
- High-dose placebo (12-17 years) (Placebo Comparator): three doses of high-dose placebo at the schedule of day 0, 21，42.
  Interventions: Other: Placebo control

INTERVENTIONS:
Biological: Recombinant COVID-19 vaccine (Sf9 cells) — This vaccine is made by using baculovirus as a vector and expressing SARS-CoV-2 S-RBD in Sf9 cells, which is purified
  Arms: High-dose vaccine (12-17 years); Low-dose vaccine (6-11 years); Medium-dose vaccine (12-17 years); Medium-dose vaccine (6-11 years)
Other: Placebo control — Except for the absence of study vaccine antigen, all other components (aluminum hydroxide, sodium chloride, sodium
  Arms: High-dose placebo (12-17 years); Low-dose placebo (6-11 years); Medium-dose placebo (12-17 years); Medium-dose placebo (6-11 years)

SUMMARY:
This is a phase Ⅰ/Ⅱ, single-center, randomized, double-blind, placebo-controlled study, to evaluate the safety, tolerability and immunogenicity of the recombinant COVID-19 vaccine (Sf9 cells) in the subjects from healthy aged 6-17 years with immunization procedures 0, 21, 42 days and doses (10μg/20μg/40μg).

DETAILED DESCRIPTION:
This is a phase Ⅰ/Ⅱ, single-center, randomized, double-blind, placebo-controlled study, to evaluate the safety, tolerability and immunogenicity of the recombinant COVID-19 vaccine (Sf9 cells) in the subjects from healthy aged 6-17 years with immunization procedures 0, 21, 42 days and doses (10μg/20μg/40μg). The phase Ⅰ clinical trials designed 4 research group, including immunization procedures 0, 21 42 days , three doses (10μg/0.25ml, 20μg/0.5ml, 40μg/1.0ml) and two ages group (6-11 and 12-17years): Each group including 30 participants. Vaccination or placebo group will be randomly assigned to receive in a 2:1 ratio, 120 in total. The phase Ⅱ clinical trials designed 4 research group, including immunization procedures 0, 21 42 days , three doses (10μg/0.25ml, 20μg/0.5ml, 40μg/1.0ml) and two ages group (6-11 and 12-17years): Each group including 120 participants. Vaccination or placebo group will be randomly assigned to receive in a 2:1 ratio, 480 in total.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-17 years；
* The subject and/or guardian can understand and voluntarily sign the informed consent form (double signature is required for 8-17 years old)；
* Reproductive women have a negative pregnancy test before each vaccination；
* The subjects are able and willing to comply with the requirements of the clinical trial protocol, and can complete the study follow-up for approximately 13.5 months.

Exclusion Criteria:

* History of SARS-CoV-2 infection.
* The COVID-19 antibody (IgG and IgM) screening was positive.
* History of asthma, history of allergy to vaccines or vaccine components, or severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioedema.
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Autoimmune diseases or immunodeficiency/immunosuppression.
* Severe chronic diseases that cannot be controlled by drugs, severe cardiovascular diseases, diabetes, liver and kidney diseases, malignant tumors, etc.
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness.
* Any condition caused by thyroid disease or history of thyroidectomy, hypersplenism, or splenectomy.
* Diagnosis of abnormal blood clotting function (for example, lack of clotting factors, coagulopathy, abnormal platelets) or obvious bruising or blood clotting.
* In the past 6 months, received immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding corticosteroid spray therapy for allergic rhinitis, and superficial corticosteroid therapy for acute uncomplicated dermatitis).
* Laboratory test results with clinically significant abnormalities (severity level 2 and above) (applicable to phase I clinical trials only).
* Received blood products in the last 3 months.
* Receive other study drugs or vaccines within the past 30 days.
* Vaccination against live attenuated vaccines in the past 30 days.
* Inactivated vaccine or subunit vaccine in the past 14 days.
* Acute disease or acute exacerbation of chronic disease in the last 7 days.
* Axillary temperature> 37.0°C.
* According to the judgment of the investigator, the subject has other factors that are not suitable for participating in the clinical trial.

Subsequent dose exclusion criteria:

In this trial, the second/third dose of vaccination may be stopped in some cases. This includes allergic reactions, severe hypersensitivity reactions, or grade 3 or higher adverse reactions that cannot be tolerated after previous vaccination/placebo. If these reactions occur, the subject should not continue to receive the second/third vaccination.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Phase I clinical trial：The incidence of adverse reactions (ARs) . | Day 0-7 days after each vaccination.
  Adverse reactions (ARs) in each dose group 0-7 days after each vaccination.
Phase II clinical trial：The incidence of adverse reactions (ARs) . | Day 0-7 days after each vaccination.
  Adverse reactions (ARs) in 0-7 days after each vaccination.
Phase II clinical trial：The geometric mean titer(GMT) of specific antibody. | Day 30 after completion of 3 doses vaccination
  The geometric mean titer (GMT) of the S-RBD protein-specific IgG antibody against SARS-CoV-2.
Phase II clinical trial：The geometric mean titer(GMT) of specific antibody. | Day 30 after completion of 3 doses vaccination
  The geometric mean titer (GMT) of anti-SARS-CoV-2 specific neutralizing antibody (neutralization test method for live virus and/or pseudovirus).

SECONDARY OUTCOMES:
Phase I/II clinical trial：The incidence of adverse events (AEs) | Day 0-7 days after each vaccination.
  Adverse events (AEs) in 0-7 days after each vaccination.
Phase I/II clinical trial：The incidence of adverse events (AEs) in all participants. | Day 0 to 30 days after completion of 3 doses vaccination
  The incidence of adverse events (AEs) from Day 0 through 30 days after completion of 3 doses vaccination in all participants.
Phase I/II clinical trial：The incidence of serious adverse events(SAEs) in all participants. | Day 0 to 30 days after completion of 3 doses vaccination
  The incidence of serious adverse events(SAEs) from Day 0 through 30 days after completion of 3 doses vaccination in all participants.
Phase I/II clinical trial：The incidence of serious adverse events(SAEs) in all participants. | Day 0 to 12 months after completion of 3 doses vaccination
  The incidence of serious adverse events(SAEs) from Day 0 through 12 months after completion of 3 doses vaccination in all participants.
Phase I clinical trial：Changes in laboratory test indicators | within 7 days before the first vaccination and on the 3rd day after each vaccination
  Changes in laboratory test indicators within 7 days before the first vaccination and on the 3rd day after each vaccination（Including white blood cell count, lymphocyte count, neutrophil count, platelets, hemoglobin, alanine aminotransferase ALT, aspartate aminotransferase AST, total bilirubin, fasting blood glucose, creatinine, prothrombin time, partially activated prothrombin time, urine Protein, urine red blood cells）
Phase I clinical trial：The geometric mean titer (GMT) of anti-COVID-19 S-RBD protein specific antibody | Day 14, Day 30，month 3, month 6, and month 12 after completion of 3 doses vaccination
  The geometric mean titer (GMT) of anti-COVID-19 S-RBD protein specific antibody (ELISA method) on day 14, day 30，month 3, month 6, and month 12 after completion of 3 doses vaccination.
Phase I clinical trial：The positive conversion rate of anti-COVID-19 S-RBD protein specific antibody. | Day 14, Day 30，month 3, month 6, and month 12 after completion of 3 doses vaccination
  The positive conversion rate of anti-COVID-19 S-RBD protein specific antibody (ELISA method) on day 14, day 30，month 3, month 6, and month 12 after completion of 3 doses vaccination.
Phase I clinical trial：the geometric mean increase multiple (GMI) of anti-COVID-19 S-RBD protein specific antibody. | Day 14, Day 30，month 3, month 6, and month 12 after completion of 3 doses vaccination
  the geometric mean increase multiple (GMI) anti-COVID-19 S-RBD protein specific antibody (ELISA method) on day 14, day 30，month 3, month 6, and month 12 after completion of 3 doses vaccination.
Phase I clinical trial：The geometric mean titer (GMT) / positive conversion rate/geometric mean growth multiple (GMI) of anti-COVID-19 specific neutralizing antibody | Day 14, Day 30，month 3, month 6, and month 12 after completion of 3 doses vaccination
  The geometric mean titer (GMT) / positive conversion rate/geometric mean growth multiple (GMI) of anti-COVID-19 specific neutralizing antibody (neutralization test method for live virus and/or pseudovirus) on day 14, day 30，month 3, month 6, and month 12 after completion of 3 doses vaccination.
Phase II clinical trial：The positive conversion rate/geometric mean growth multiple (GMI) of anti-COVID-19 S-RBD protein specific antibody | Day 14, Day 30, month 6, and month 12 after completion of 3 doses vaccination
  The positive conversion rate/geometric mean growth multiple (GMI) of anti-COVID-19 S-RBD protein specific antibody on day 14, Day 30, month 6, and month 12 after completion of 3 doses vaccination
Phase II clinical trial：The positive conversion rate/geometric mean growth multiple (GMI) of anti-COVID-19 specific neutralizing antibody | Day 14, Day 30, month 6, and month 12 after completion of 3 doses vaccination
  The positive conversion rate/geometric mean growth multiple (GMI) of anti-COVID-19 specific neutralizing antibody (neutralization test method for live virus and/or pseudovirus) on day 14, day 30，month 3, month 6, and month 12 after completion of 3 doses vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China